CLINICAL TRIAL: NCT03892486
Title: Analysis of the Effect of a Diet Enriched With Polyunsaturated Fatty Acids on the Proteomic and Metabolomic Profiles of Blood Plasma of Healthy People Aged 18-50
Brief Title: Polyunsaturated Fatty Acids Supplementation and Blood Metabolome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: LKB 1249/19
Record Dates: First submitted 2019-02-21; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: metabolomics, proteomics, PUFA, nutrition; healthy people aged 18-50

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The high PUFA diet group (Experimental): This will receive detailed nutritional recommendations and will consume at least 4 table spoons of olive oil or 30 grams of nuts daily for 12 weeks.
  Interventions: Other: The high PUFA diet group
- Control group (No Intervention): The Control group will receive general nutritional recommendations based on Human Nutrition Recommendations for Polish Population.

INTERVENTIONS:
Other: The high PUFA diet group — Assumptions of nutritional intervention: in a randomized manner volunteers will be assigned to one of two groups: a control group which will receive general nutritional recommendations, based on the Polish nutrition pyramid, and the intervention group which will receive nutritional recommendations, based on the Polish nutrition pyramid and will consume at least 4 tablespoons of olive oil or 30 grams of nuts every day for 12 weeks.
  Arms: The high PUFA diet group

SUMMARY:
Analysis of the effect of dietary intervention based on increased polyunsaturated fatty acid intake on health. Specifically changes in blood lipid profile, as well as proteomic and metabolomic profiles of healthy adults will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* good health,
* proper body weight
* not meeting the needs for polyunsaturated fatty acids

Exclusion Criteria:

* increased body weight,
* limited communication to an extent that makes it impossible to carry out a food interview,
* eating disorders (according to food history),
* metabolic diseases,
* pregnancy,
* lactation,
* taking drugs that influence the metabolism of lipids or carbohydrates

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Nutrient intake | 12 weeks
  Nutrient intake (3-day food records)
Concentrations of lipoproteins and glucose | 12 weeks
  Serum concentrations of lipoproteins and glucose at baseline and after the intervention [mg/dl]
Proteomic analysis of plasma | 12 weeks
  The aim is to identify biomarkers in the blood and to determine the differences between people from the control and the intervention group
Metabolite concentrations in plasma | 12 weeks
  Metabolite concentrations in plasma samples are measured by high resolution mass spectrometry at baseline and after the intervention

SECONDARY OUTCOMES:
Body mass | 12 weeks
  body mass at baseline and after the intervention
Height | 12 weeks
  height
Percentage body fat | 12 weeks
  percentage body fat at baseline and after the intervention
Waist circumference | 12 weeks
  waist circumference at baseline and after the intervention
hip circumference | 12 weeks
  hip circumference at baseline and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Agata Chmurzynska, PhD, Principal Investigator — Poznan University of Life Sciences
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland